CLINICAL TRIAL: NCT00782925
Title: An Educational and Exercise Program as Secondary Prevention of Recurrent Lower Back Pain in Healthcare Workers: A Randomized, Controlled, 2-year Follow-up Study.
Brief Title: An Educational and Exercise Program as Secondary Prevention of Recurrent Lower Back Pain in Healthcare Workers
Acronym: PRESLO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2008.511
Record Dates: First submitted 2008-10-30; First posted 2008-10-31 (Estimated); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Acute Low Back Pain
Keywords: Low back pain; recurrence; chronic low back pain; educational program; physical therapy; home exercise; compliance
MeSH Terms: conditions — Low Back Pain; Recurrence; Patient Compliance | interventions — Resistance Training

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Study intervention:
  * A face/profile X-ray of their entire spine at baseline
  * Educational program
  * Exercise program
  * Self-led exercises
  * A follow-up at 12 and 24 months with their occupational therapist.
  * A follow-up at 18 months with a physical therapist.
  * Workers received also at the end of the educational program written standardized information about back pain ("the back book", an information booklet) 1.
    1. Coudeyre E., Tubach F., Rannou F. & all, Effect of simple information booklet on pain persistance after an acute episode of low back pain: a non- randomised trial in a primary care setting. PLoS ONE. 2007 ; 2 : e706
  Interventions: Other: educational program; Other: exercise program; Other: Self-led exercises
- 2 (No Intervention): Control intervention :
  * No intervention
  * A face/profile X-ray of their entire spine at baseline
  * A follow-up at 12 and 24 months with their occupational therapist,
  * A follow-up at 18 months with a physical therapist.

INTERVENTIONS:
Other: educational program — Educational program will consist of 1, 2-hour, small-group (8-patient) session with a specialist physician in Physical and Rehablilitation Medecine. Workers will be given information about lower back pain, pain and psychosocial risk factors for persistent or recurrent back-related disability
  Arms: 1
Other: exercise program — The exercise program will consist of 5, 90-minute, small-group (8-patient) sessions with a physical therapist. Healthcare workers will be taught exercises including warm-ups, floor exercises, and endurance training. Only one absence will be allowed, otherwise the worker will be considered as non-compliant.
  Arms: 1
Other: Self-led exercises — Self-led exercises to perform as part of a daily exercise routine
  Arms: 1

SUMMARY:
At Lyon University Medical Center, back problems are the leading cause of sick leave. The course of lower back pain is usually relatively short (recovery occurs within 4 to 6 weeks in 90% of cases). However, about 5-10% develop chronic lower back pain. Although this is a relatively small group, the economic consequences are enormous (accounting for 70 to 80% of the total cost of lower back pain).

Nowadays, some very general training sessions are offered to workers at Lyon University Medical Center, irrespective of their lower back pain status. These very general training sessions are mostly preventive and primary in nature (like back school program) despite the fact that these people already have a history of lower back pain, the main risk factor of recurrence and chronic pain.

Since the 1980, some multidisciplinary functional restoration programs have been advised as a strategy for secondary and tertiary prevention of lower back pain.

The purpose of this randomized controlled trial is to assess the effectiveness of physical exercise combined with an educational program and self-led exercise for Lyon University Medical Center workers with lower back pain. We hope this intervention will reduce the risk of recurrence and chronic lower back pain.

ELIGIBILITY:
Inclusion Criteria:

* All healthcare workers in the 4 hospital sites
* History of acute or subacute lower back pain in the 3 past years

Exclusion Criteria:

* History of surgery for spinal fractures
* History of lumbosacral arthrodesis
* History of surgical intervention or discal hernia, more than 2 levels or more than twice
* Radiculalgia with sign of motor deficit, or radiculalgia with a positive Lasègue sign
* Eligible for enrollement in a functional restoration program for lower back pain
* Ongoing low back pain (lumbago)
* Psychosocial or behavioural impairment
* Unstable cardiac disease
* Inability to fill out the questionnaires and scales (inability to understand French)
* Pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 351 (Actual)
Dates: Start 2008-10; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Percentage of patients with recurrence(s) of lower back pain (number of related days of sick leave) over 12 months and 24 months | 12 and 24 months

SECONDARY OUTCOMES:
Recurrences of lower back pain | At baseline, 12 and 24 months after intervention
Delay before a recurrence of lower back pain | At baseline, 12 and 24 months after intervention
Percentage of patients with a chronic lower back pain (sick leave days>3 months) | At baseline, 12 and 24 months after intervention
Lower back function | At baseline, 12 and 24 months after intervention
Pain : characteristics, intensity (Quebec Back Pain Disability Scale) | At baseline, 12 and 24 months after intervention
Fear-avoidance beliefs(FABQ scale) | At baseline, 12 and 24 months after intervention
Quality of life (SF-12 scale) | At baseline, 12 and 24 months after intervention
Depression and anxiety (HAD scale) | At baseline, 12 and 24 months after intervention
Participant compliance with the global prevention program (self-led exercises) | At 6 and 12 months after intervention
sagittal alignement of the spine (X-ray) | At baseline

CONTACTS AND LOCATIONS:
Overall Officials: Alain BERGERET, Pr, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Hospices Civils de Lyon, Lyon, France

REFERENCES:
- [Result] Denis A, Zelmar A, Le Pogam MA, Chaleat-Valayer E, Bergeret A, Colin C. The PRESLO study: evaluation of a global secondary low back pain prevention program for health care personnel in a hospital setting. Multicenter, randomized intervention trial. BMC Musculoskelet Disord. 2012 Nov 27;13:234. doi: 10.1186/1471-2474-13-234. PMID 23181446
- [Result] Chaleat-Valayer E, Denis A, Abelin-Genevois K, Zelmar A, Siani-Trebern F, Touzet S, Bergeret A, Colin C, Fassier JB. Long-term effectiveness of an educational and physical intervention for preventing low-back pain recurrence: a randomized controlled trial. Scand J Work Environ Health. 2016 Jun 1;42(6):510-519. doi: 10.5271/sjweh.3597. Epub 2016 Oct 3. PMID 27779639